CLINICAL TRIAL: NCT02404792
Title: Exercise for Healthy Aging: The Impact of HIV and Aging on Physical Function and the Somatopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-2207; K23AG050260 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-04-01 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: HIV; Inflammation; Obesity; Aging, Biological
Keywords: Frail Elderly; IGF-1
MeSH Terms: conditions — Inflammation; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-uninfected (Active Comparator): HIV-uninfected men and women, age 50-70 years. All participants will exercise at a moderate intensity (cardiovascular + resistance training) for 12 weeks, then will be randomized to continue moderate intensity or advance to high intensity exercise for an additional 12 weeks.
  Interventions: Other: High-intensity cardiovascular and resistance exercise; Other: Moderate-intensity cardiovascular and resistance exercise
- HIV-infected (Experimental): HIV-infected men and women, age 50-70 years. All participants will exercise at a moderate intensity (cardiovascular + resistance training) for 12 weeks, then will be randomized to continue moderate intensity or advance to high intensity exercise for an additional 12 weeks.
  Interventions: Other: High-intensity cardiovascular and resistance exercise; Other: Moderate-intensity cardiovascular and resistance exercise

INTERVENTIONS:
Other: High-intensity cardiovascular and resistance exercise
Other: Moderate-intensity cardiovascular and resistance exercise

SUMMARY:
The primary objective of this proposal is to compare a moderate or high intensity exercise intervention to improve physical function in persons aging with Human Immunodeficiency Virus (HIV).

DETAILED DESCRIPTION:
The primary objective of this proposal is to compare a moderate or high intensity exercise intervention to improve physical function in persons aging with HIV. Both HIV-infected and HIV-uninfected older adults will be assigned to a moderate intensity cardiovascular and resistance training intervention for 12 weeks, and then randomized to either continue moderate intensity exercise, or increase to high intensity exercise for an additional 12 weeks. The primary outcome is the impact of exercise on physical function, as measured by the overall score of a modified Short Physical Performance Battery (mSPPB) and the chair rise time from the mSPPB. The secondary outcomes include changes in insulin-like growth factor-1 (systemic and local) and inflammation (interleukin-6 (IL-6), soluble tumor necrosis factor receptors 1 and 2 (sTNFR-1 and sTNFR-2)).

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-75
* HIV+ must be on ART for a minimum of 2 years with viral load <200 copies/mL
* Sedentary
* cluster of differentiation 4 (CD4) T-cell count >200 cells/microliter
* BMI >19 and <41
* Among females, must be post-menopausal
* Able to perform activities of daily living with out assistance

Exclusion Criteria:

* Diabetes, poorly controlled with HgbA1c >7.5; on insulin
* On growth hormone (or growth hormone axis) therapy, intramuscular testosterone, corticosteroids.
* Known active hepatitis B or C (viremia).
* Severe liver disease
* Uncontrolled hypertension (SPB >180 or diastolic >100).
* Underlying cardiac conditions that would make exercise or exercise testing potentially unsafe (unstable ischemic heart disease, Class III or IV heart failure clinically significant aortic stenosis, uncontrolled angina, or uncontrolled arrhythmia)
* pulmonary disease requiring the use of supplemental oxygen ≥ 4 liters with physical exertion
* current diagnosis of malignancy (excluding non-melanoma skin cancers) within 48 weeks prior to enrollment
* surgery/trauma/injury/fracture within 24 weeks prior to enrollment that may impact a subject's ability to exercise
* history of stroke with residual deficits that may impact ability to exercise; orthopedic problems (e.g., severe osteoarthritis, rheumatoid arthritis) that greatly limit the ability to perform moderate-intensity resistance exercise (e.g., unable to be properly positioned in exercise equipment or to have severely restricted range of motion even after modifications have been made)
* weight over 300 pounds
* Montreal Cognitive Assessment (MOCA) score < 18 (will be evaluated at screening visit after consent obtained)
* AIDS-defining opportunistic infection within the 24 weeks prior to enrollment
* Person who appear to have unstable health, are incapable of safely participating in the exercise intervention, or are felt to have a life expectancy of < 1 year.
* Participants on anticoagulants (clopidogrel, Coumadin, etc) will be excluded from the muscle biopsy.
* Aspirin and Non-steroidal anti-inflammatory agents are not exclusions but should be stopped 1 week prior to muscle biopsy (subset of subjects).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10-02 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Erlandson, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado- Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kulik GL, Wilson MP, Jankowski CM, Fourman LT, Erlandson KM. Examining the Heterogeneity of Exercise Response Among Sedentary Older Adults: A Descriptive Analysis. J Aging Res. 2025 Mar 18;2025:6952002. doi: 10.1155/jare/6952002. eCollection 2025. PMID 40134456
- [Derived] Bowman ER, Wilson M, Riedl KM, MaWhinney S, Jankowski CM, Funderburg NT, Erlandson KM. Lipidome Alterations with Exercise Among People With and Without HIV: An Exploratory Study. AIDS Res Hum Retroviruses. 2022 Jul;38(7):544-551. doi: 10.1089/AID.2021.0154. Epub 2022 Apr 21. PMID 35302400
- [Derived] Erlandson KM, Liu J, Johnson R, Dillon S, Jankowski CM, Kroehl M, Robertson CE, Frank DN, Tuncil Y, Higgins J, Hamaker B, Wilson CC. An exercise intervention alters stool microbiota and metabolites among older, sedentary adults. Ther Adv Infect Dis. 2021 Jun 25;8:20499361211027067. doi: 10.1177/20499361211027067. eCollection 2021 Jan-Dec. PMID 34262758
- [Derived] Jankowski CM, Wilson MP, MaWhinney S, Reusch J, Knaub L, Hull S, Erlandson KM. Blunted Muscle Mitochondrial Responses to Exercise Training in Older Adults With HIV. J Infect Dis. 2021 Aug 16;224(4):679-683. doi: 10.1093/infdis/jiaa799. PMID 33378424
- [Derived] Erlandson KM, Wilson MP, MaWhinney S, Rapaport E, Liu J, Wilson CC, Rahkola JT, Janoff EN, Brown TT, Campbell TB, Jankowski CM. The Impact of Moderate or High-Intensity Combined Exercise on Systemic Inflammation Among Older Persons With and Without HIV. J Infect Dis. 2021 Apr 8;223(7):1161-1170. doi: 10.1093/infdis/jiaa494. PMID 32779711
- [Derived] Johs NA, Kellar-Guenther Y, Jankowski CM, Neff H, Erlandson KM. A qualitative focus group study of perceived barriers and benefits to exercise by self-described exercise status among older adults living with HIV. BMJ Open. 2019 Mar 7;9(3):e026294. doi: 10.1136/bmjopen-2018-026294. PMID 30850416

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With HIV: All participants were aged 50 to 75 years, sedentary (<60 minutes of physical activity each week for 6 months preceding by self-report), had a body mass index (BMI) between 20 and 40 kg/m2, and had no contraindications to initiating an exercise regimen (e.g., severe mobility limitation, unstable angina, supplemental oxygen requirement, uncontrolled hypertension). Participants with diabetes had hemoglobin A1c of 7.5% or less; sex hormone supplementation was restricted to stable, physiologic doses for ≥3 months prior to study entry and intramuscular testosterone was excluded. PLWH were on stable ART with an undetectable HIV-1 RNA for >2 years and a CD4 T-cell count >200 cells/µL. At week 12, VO2 max measurements were repeated and participants were randomized to either continue moderate-intensity exercise or advance to high-intensity (60-70% of week 13 VO2 max and >80% 1-RM) for the remaining 12 weeks.
- HIV-Uninfected Controls: All participants were aged 50 to 75 years, sedentary (<60 minutes of physical activity each week for 6 months preceding by self-report), had a body mass index (BMI) between 20 and 40 kg/m2, and had no contraindications to initiating an exercise regimen (e.g., severe mobility limitation, unstable angina, supplemental oxygen requirement, uncontrolled hypertension). Participants with diabetes had hemoglobin A1c of 7.5% or less; sex hormone supplementation was restricted to stable, physiologic doses for ≥3 months prior to study entry and intramuscular testosterone was excluded.At week 12, VO2 max measurements were repeated and participants were randomized to either continue moderate-intensity exercise or advance to high-intensity (60-70% of week 13 VO2 max and >80% 1-RM) for the remaining 12 weeks.
Period: Overall Study
Arm/Group | Participants With HIV | HIV-Uninfected Controls
Started | 32 | 37
Completed | 27 | 29
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- HIV-Uninfected Controls: All participants were aged 50 to 75 years, sedentary (<60 minutes of physical activity each week for 6 months preceding by self-report), had a body mass index (BMI) between 20 and 40 kg/m2, and had no contraindications to initiating an exercise regimen (e.g., severe mobility limitation, unstable angina, supplemental oxygen requirement, uncontrolled hypertension). Participants with diabetes had hemoglobin A1c of 7.5% or less; sex hormone supplementation was restricted to stable, physiologic doses for ≥3 months prior to study entry and intramuscular testosterone was excluded. PLWH were on stable ART with an undetectable HIV-1 RNA for >2 years and a CD4 T-cell count >200 cells/µL.
  At week 12, VO2 max measurements were repeated and participants were randomized to either continue moderate-intensity exercise (40-50% VO2 max and 60-70% 1-RM) or advance to high-intensity (60-70% of week 13 VO2 max and >80% 1-RM) for the remaining 12 weeks.
- Participants With HIV: All participants were aged 50 to 75 years, sedentary (<60 minutes of physical activity each week for 6 months preceding by self-report), had a body mass index (BMI) between 20 and 40 kg/m2, and had no contraindications to initiating an exercise regimen (e.g., severe mobility limitation, unstable angina, supplemental oxygen requirement, uncontrolled hypertension). Participants with diabetes had hemoglobin A1c of 7.5% or less; sex hormone supplementation was restricted to stable, physiologic doses for ≥3 months prior to study entry and intramuscular testosterone was excluded. PLWH were on stable ART with an undetectable HIV-1 RNA for >2 years and a CD4 T-cell count >200 cells/µL.
  At week 12, VO2 max measurements were repeated and participants were randomized to either continue moderate-intensity exercise (40-50% VO2 max and 60-70% 1-RM) advance to high-intensity (60-70% of week 13 VO2 max and >80% 1-RM) for the remaining 12 weeks.
- Total: Total of all reporting groups
Arm/Group | HIV-Uninfected Controls | Participants With HIV | Total
Number analyzed (Participants) | 37 | 32 | 69
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 58.7 (6.9) | 56.8 (5.7) | 57.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 35 | 28 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 33 | 28 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 9 | 12
  White | 31 | 20 | 51
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Rise From a Chair 10 Times (Modified From the Original Short Physical Performance Battery)
Description: Chair rise time is measured as a continuous variable of time to stand up from a sitting position 10 times. Lower number = faster; larger number = slower
Time Frame: 24 weeks
Population: 37 and 32 had baseline values; 29 and 27 (uninfected and with HIV, respectively) completed 24 weeks.
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | HIV-uninfected Controls | Participants With HIV
Number analyzed (Participants) | 37 | 32
percentage change
  Change 0-12 weeks: number analyzed (Participants) | 31 | 28
  Change 0-12 weeks | -20 [-24 to -16] | -20 [-24 to -16]
  Change 13-24 weeks: number analyzed (Participants) | 29 | 27
  Change 13-24 weeks | -8 [-12 to -4] | -10 [-14 to -5]

2. Secondary Outcome: Changes in Insulin-like Growth Factor (IGF)-1
Description: Measures at baseline and following 24 weeks of exercise
Time Frame: 24 weeks
Population: Missing data on one participant with HIV that completed the study. Data listed below ONLY includes data on persons with measurements at both baseline and week 24.
Measure: Geometric Mean (95% Confidence Interval); unit: IGF-1 (ng/mL)
Arm/Group | Participants With HIV | HIV-Uninfected Controls
Number analyzed (Participants) | 26 | 29
IGF-1 (ng/mL)
  Baseline | 79.87 [66.33 to 96.18] | 86.4 [78.46 to 95.13]
  Week 24 | 85.42 [69.49 to 104.99] | 84.65 [76.77 to 93.34]

3. Secondary Outcome: Changes in Inflammation (Interleukin-6 [IL-6], Soluble Tumor Necrosis Factor Receptors 1 and TNF-alpha.
Description: The primary outcome is change from 0 to 24 weeks. These changes in inflammation are measured at baseline (pre-exercise) and at 24 weeks (post exercise).
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | HIV-uninfected Controls | Participants With HIV
Number analyzed (Participants) | 37 | 32
percentage of change
  Change in IL-6 | -2 [-16 to 22] | 10 [-10 to 34]
  Change in sTNFr1 | 2.3 [-3.5 to 8.3] | -2.5 [-8.2 to 3.6]
  Change in TNFalpha | 1.3 [-11.1 to 15.4] | -2.5 [-15 to 11.7]

ADVERSE EVENTS:
Time Frame: Adverse data were collected up at each study visit for up to 24 weeks through completion of the exercise intervention, and for 3 days following muscle biopsy, in participants who received a biopsy following completion of the exercise intervention.
Description: Events were described as definite, probable, or possible in relation to the exercise intervention or related to other study procedures. Participants reported any AE in real-time. Additionally, participants completed a health information sheet every 2-3 weeks where they were asked about any calls or visits to their provider, hospitalizations, or imaging.
Arm/Group | HIV-uninfected Controls | Participants With HIV
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 9/37 | 17/32
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-uninfected Controls (N=37) | Participants With HIV (N=32)
Musculoskeletal injury/pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 13 (20) — Included aches, pains, strains, etc.
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizzyness or lightheadedness (Cardiac disorders) | 0 (0) | 4 (4)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) — Pre, post, or during exercise
Chest pain and shortness of breath (Cardiac disorders) | 1 (1) | 0 (0) — Minor, resolved with rest
Fatigue (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02404792/Prot_SAP_000.pdf